CLINICAL TRIAL: NCT07375784
Title: UP-GRADE: Assessment Pathways for Psychopathological Aspects and Psychological Support in the Adolescent Population (UG) A Prospective, Single-center, Longitudinal Study of Pediatric Patients Aged 14 to 17 Years With Psycho-relational Distress Treated at the Pediatric Department of the Policlinico San Matteo in Pavia.
Brief Title: UP-GRADE: Assessment Pathways for Psychopathological Aspects and Psychological Support in the Adolescent Population
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Amelia Licari, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: UP-GRADE
Record Dates: First submitted 2025-12-31; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Psychological Distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Q-PAD questionnaire — The Q-PAD is a questionnaire designed to assess psychopathology in adolescence, measure the level of adjustment, and evaluate overall well-being.
  The minor will be presented with statements and asked to indicate their response using a scale from 1 (the statement is false/does not describe my situation or opinion at all) to 4 (the statement is true/accurately describes my situation or opinion). This questionnaire has been validated on a sample of 1,454 individuals aged between 14 and 19 years and is used to investigate anxiety, depression, body dissatisfaction, substance abuse, interpersonal conflicts, family problems, uncertainty about the future, psychosocial risk, self-esteem, and well-being.
  The questionnaire is evaluated at 3 different time points during the study: at T0 and at T1 (+6 months).

SUMMARY:
The objective of the observational study "UP-GRADE: Assessment of Psychopathological Aspects and Psychological Support in the Adolescent Age Group of the Population. A Monocentric Longitudinal Interventional Study with Prospective Enrollment of Pediatric Patients Aged 14-17 with Psychosocial Distress in the Pediatric Department of the Policlinico San Matteo in Pavia" is to explore the psycho-emotional state of a sample of adolescents aged 14-17 in a population of patients under the care of the Pediatric Unit, at the Fondazione IRCCS Policlinico San Matteo. The study aims to estimate the proportion of subjects with altered anxiety levels (compared to the reference population). A secondary objective is to estimate the proportion of subjects with distress levels (compared to the reference population) in other psychosocial areas, based on the Q-PAD questionnaire score. Additionally, for patients with altered scores in at least one subscale of the Q-PAD, the study will assess the effect of a psychological support program consisting of 10 counseling sessions.

The subjects involved in the study must meet the following inclusion criteria: being aged between 14 and 17 at the time of enrollment, having access to hospital services, having exhibited psychosocial distress, understanding the Italian language, and signing informed consent. Finally, it is specified that the study does not involve any interventions or potentially invasive instrumental investigations.

DETAILED DESCRIPTION:
The protocol is structured in two phases: an initial screening meeting and the follow-up of each participant through 10 psychological support sessions.The follow-up will consist of 10 psychological support sessions, each lasting 1 hour, at a biweekly interval. It is specified that during the second meeting, the Q-PAD questionnaire-used for the evaluation of psychopathology in adolescence-will be administered. Finally, a retest with the same questionnaire will be conducted at the end of the last psychological support session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 17 years
* Access to hospital services
* Manifestation of psychological distress
* Understanding the Italian language
* Signing of informed consent

Exclusion Criteria:

* Age <14 years or ≥18 years at enrollment

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample will consist of 80 subjects under the care of the Pediatric Unit, Policlinico San Matteo, Pavia, considering the prospective recruitment of patients who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Q-PAD questionnaire score at T0 | Baseline-day 1. The term T0 refers to the baseline visit, the first visit planned in the schedule of activities.
  Estimate the proportion of subjects with altered anxiety levels (compared to the reference population) using the Q-PAD questionnaire. The assessment is at T0.

SECONDARY OUTCOMES:
Assessment of psychological distress in patients with altered values detected using the Q-PAD questionnaire | Between T0 and T1. The term T0 refers to the baseline visit, that is, the first visit scheduled in the schedule of study activities and the term T1 refers to the last visit scheduled according to the protocol procedures (visit 10-after six months).
  Estimate the proportion of subjects with distress levels (compared to the reference population) in other psychosocial areas and assess, in the group of patients with altered values in at least one subscale of the Q-PAD, the effect of a 10-session psychological support program.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Pediatria, Pavia, Pavia, Italy